CLINICAL TRIAL: NCT06790433
Title: Comparison Between the Dentapen and Vibraject: a Randomized Clinical Study on the Administration of Local Anaesthesia in Adult Patients.
Brief Title: Comparison Between the Dentapen and Vibraject
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riyadh Elm University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dr Ammar's - Anesthesia 2025
Record Dates: First submitted 2025-01-09; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Pain
Keywords: dental injection
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibraject (Active Comparator): Participants will receive dental injection using Vibraject
  Interventions: Device: Vibraject
- Dentapen (Active Comparator): Participants will receive dental injection using Dentapen
  Interventions: Device: Dentapen

INTERVENTIONS:
Device: Vibraject — The needle was advanced into the tissue until it was estimated to be over the root apex while remaining parallel to the tooth's long axis. The Vibraject was activated after aspiration to deposit the solution slowly at approximately 50 seconds. Following cartridge deposition, the operator adjusted the participant to an upright seated position
  Arms: Vibraject
Device: Dentapen — The needle was advanced into the tissue until it was estimated to be over the root apex while remaining parallel to the tooth's long axis (needle placement). The Dentapen was activated after aspiration to deposit the solution at a medium rate (1 mL/60 s) using the ramp-up mode. Following cartridge deposition, the operator adjusted the participant to an upright seated position
  Arms: Dentapen

SUMMARY:
A split-mouth, controlled trial aimed to assess patient-reported pain levels during local anaesthesia administration to the buccal side of the maxillary posterior teeth using Vibraject-assisted injection and the Dentapen® system in its ramp-up mode.

Pain intensity was evaluated using the Visual Analogue Scale immediately following each injection, and heart rate measurements were recorded before and after each injection. Patient preferences for injection methods were also documented

DETAILED DESCRIPTION:
Steps of the Experiment

The experimental protocol was meticulously structured to evaluate the efficacy and patient response to two different local anaesthetic delivery systems. The steps were as follows:

Step I: Before administering a local anaesthetic, the patient's heart rate was checked with a pulse oximeter (Beurer Finger Pulse Oximeter). The results were recorded.

Step II: Patients were randomly assigned to get the injection of local anaesthetic at their initial appointment either with the Dentapen system (ramp-up) or with Vibraject. To simplify the protocol, a 27-gauge needle was used for all dental injections with bevel side directly headed to the injected site.

Step III: In the next appointment, after of one hour on a digital timer, the other technique was used for the same patients on the other side. Hence, each patient was given local anaesthesia twice, once with the Dentapen system (ramp-up mode) and once with Vibraject.

Step IV: Immediately after each local anesthesia injection operation, the patient was asked to use the Visual Analogue Scale to score the intensity of reported pain.

Step V: After administering a local anaesthetic, the patient's heart rate was measured with a pulse oximeter (Beurer Finger Pulse Oximeter). The results were recorded.

Step VI: After both injections were administered to each patient, they were asked which injection they would prefer by selecting the injection number (first or second) according to their order for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Individuals classified under American Society of Anesthesiologists classes I and II, indicating a healthy or mild systemic disease status.
* Individuals aged from 18 up to 65 years, encompassing both male and female patients.
* Individuals who required local anesthetic injections bilaterally in the buccal side of the upper posterior teeth. These injections were necessary for various dental procedures, including restorative, endodontic, or prosthodontic treatments, and volunteers as well were to be administered across both sides of upper posterior teeth.
* Individuals must be in good health, not currently taking any medication, and have no contraindications to the use of local anesthesia.
* Individuals who have the ability to understand both oral and written instructions, ensuring effective communication and comprehension throughout the study.

Exclusion Criteria:

* Individuals with allergies to local anesthetics, this is to prevent adverse reactions.
* Pregnant or nursing women, this is to avoid any potential risks to their health or that of their infants.
* Individuals who were actively taking drugs that could alter pain perception or anxiety levels, such as nonsteroidal anti-inflammatory drugs, opioids, or antidepressants. This was to ensure that the study's findings on pain perception were not influenced by external substances
* Individuals with heavy alcohol consumption. .
* Patients with active pathologies at the injection site, this is to avoid complications and to ensure the accuracy of the study's results.
* Individuals who could not commit to the study's schedule or were unable to give informed consent. This ensured that all participants were fully aware of and agreeable to the study's procedures and requirements.
* Patients who required intravenous sedation for their dental procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Heart rate | Immediately after the intervention/procedure (dental anesthesia)
  Heart rate was measured for the participants using a pulse oximeter
Pain rating scale | 3 minutes after the intervention/procedure (dental anesthesia)
  After each local anesthesia injection operation, the patient was asked to use the Visual Analogue Scale to score the intensity of reported pain. It is a scale of pain composed of 10 scores from 0 to 10, a higher score indicates greater pain intensity (worse outcome).
Participant's future preference | 5 minutes after the intervention/procedure (dental anesthesia)
  The participants were asked using a simple questionnaire to state their preference for the delivery system of future injections

CONTACTS AND LOCATIONS:
Overall Officials: ِAmmar AbuMostafa, MSc, Study Director — Riyadh Elm University
Locations (1):
- Dental Hospitals - Riyadh Elm University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-01-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT06790433/Prot_SAP_ICF_000.pdf